CLINICAL TRIAL: NCT06999252
Title: The Combination of Rimegepant and PD-1 Inhibitor in the Treatment of Liver Metastasis Colorectal Cancer
Brief Title: Rimegepant Combined With PD-1 in Liver Metastasis Colorectal Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Li Dawei, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Passion CRC
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — rimegepant sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients will be treated with Rimegepant and PD-1 (Experimental)
  Interventions: Drug: Rimegepant; Drug: PD-1

INTERVENTIONS:
Drug: Rimegepant — Take 75 mg every other day
Drug: PD-1 — 200mg intravenously every 3 weeks (Q3W), was administered until the occurrence of unacceptable toxic effects, or disease progression, withdrawal of consent, or withdrawal as judged by the investigator.

SUMMARY:
The goal of this clinical trial is to learn about efficacy of Rimegepant in combination with PD-1 in patients with liver metastasis colorectal cancer. The main question is to explore the survival time, safety and tolerability of the treatment. At the same time, the correlation between biomarkers (including PD-L1 expression, tumor mutation load, lymphocyte subpopulation, cytokines, TCR, intestinal microbes, and others) and the efficacy and drug resistance mechanism will be analyzed, so as to provide reference for the subsequent guidance of the screening of benefit groups.

ELIGIBILITY:
* Inclusion Criteria:

  1. Age ≥18 years old, both sexes ;
  2. Patients with histologically or cytologically confirmed locally advanced and advanced colorectal cancer that cannot be R0 resected;
  3. Recist1.1-defined disease progression or intolerance to prior standard therapy during or after standard therapy. Standard therapy was required to include all the following agents: fluorouracilines, chemotherapy agents such as irinotecan, and oxaliplatin, with or without an anti-VEGF monoclonal antibody (e.g., bevacizumab). Left-sided KRAS/NRAS/BRAF wild-type subjects received combined anti-EGFR mAb (cetuximab or panitumumab).

  5. Patients with ECOG score of 0-1 and expected survival time ≥3 months, patients who can cooperate to observe adverse reactions and efficacy; 6. At least one measurable tumor lesion according to RECIST 1.1 criteria; 7. Good organ function:
  1. neutrophil ≥1.5*109/L; Platelet ≥100*109/L; Hemoglobin ≥9g/dl; Serum albumin ≥3g/dl;
  2. Thyroid stimulating hormone (TSH) ≤ 1 times the upper limit of normal, T3 and T4 in the normal range;
  3. bilirubin ≤ 1.5 times the upper limit of normal value; ALT and AST≤ 2 times the upper limit of normal;
  4. Serum creatinine ≤ 1.5 times the upper limit of normal, creatinine clearance ≥60ml/min;
  5. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times the upper limit of the normal range, unless the patient is receiving anticoagulant therapy and the PT value is within the intended range for anticoagulant therapy;
  6. Activated partial thromboplastin time (aPTT) ≤ 1.5 times the upper limit of normal; 8. There were no serious concomitant diseases that could make the survival time less than 5 years; 9. Negative pregnancy test in female subjects (for female patients of childbearing potential); Infertile female patients; 10. Male patients of childbearing potential and female patients of childbearing potential and at risk of pregnancy must agree to use adequate contraception for the entire duration of the study and for 12 months after receiving treatment with the protocol; 11. Signed and dated informed consent indicating that the patient has been informed about all relevant aspects of the study; 12. Patients who are willing and able to comply with the visit schedule, treatment plan, laboratory tests, and other study procedures; 13. Willing to comply with the arrangement during the study period can not participate in any other clinical research on drugs and medical devices.

Exclusion Criteria:

1. Pathological diagnosis of other intestinal tumors, such as gastrointestinal stromal tumor;
2. Prior treatment with PD-1 antibody;
3. Prior treatment with mTOR inhibitor;
4. Previous or concurrent history of other malignant tumors, excluding adequately treated non-melanoma skin cancer, cervical carcinoma in situ and thyroid papillary carcinoma;
5. Active autoimmune disease, history of autoimmune disease (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); It does not include autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes on stable doses of insulin; Vitiligo or cured childhood asthma/allergy without any intervention in adulthood;
6. A history of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation or allogeneic bone marrow transplantation;
7. Contraindications to antiangiogenic drugs (such as active bleeding, gastrointestinal bleeding, hemoptysis, etc.);
8. History of interstitial lung disease (excluding radiation pneumonitis without steroid treatment) and non-infectious pneumonia;
9. Patients with active pulmonary tuberculosis infection detected by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or with a history of active pulmonary tuberculosis infection more than 1 year before enrollment but without regular treatment;
10. The subject has active hepatitis B (HBV DNA ≥2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive and HCV-RNA above the detection limit of the assay)
11. Severe cardiopulmonary and renal dysfunction;
12. Have hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
13. A history of psychotropic substance abuse, alcohol or drug abuse;
14. Other factors that may affect subject safety or trial compliance as judged by the investigator. Severe medical conditions requiring concomitant treatment (including mental illness), serious laboratory abnormalities, or other family or social factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 2 year

SECONDARY OUTCOMES:
progression-free survival (PFS） | 2 years
overall survival (OS) | 4 years
disease control rate (DCRs) | 2 years
advert events | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No